CLINICAL TRIAL: NCT03766477
Title: Aspects Associated With Bruxism and Sleep Quality
Brief Title: Aspects Associated With Sleep Quality
Status: Completed | Type: Observational
Sponsor: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, Noéli Boscato, PhD, Associate Professor, Federal University of Pelotas
Other Study IDs: FUPelotas2
Record Dates: First submitted 2018-11-06; First posted 2018-12-06 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Sleep Bruxism
Keywords: Sleep bruxism; Sleep; Sleep hygiene
MeSH Terms: conditions — Sleep Bruxism; Sleep Hygiene | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals with sleep bruxism: Individuals with sleep bruxism evaluated in three different methods regarding their sleep quality:
  * Pittsburgh Sleep Quality Index (IQSP) and Johansson
  * Smartphone APP
  * Polysomnography
  Interventions: Diagnostic Test: Pittsburgh Sleep Quality Index (IQSP) and Johansson; Diagnostic Test: Smartphone APP; Diagnostic Test: Polysomnography

INTERVENTIONS:
Diagnostic Test: Pittsburgh Sleep Quality Index (IQSP) and Johansson — All participants will to answer the Pittsburgh Sleep Quality Index (IQSP) and Johansson questionnaires before polysomnography examination and use of APP.
Diagnostic Test: Smartphone APP — All study participants will use a smartphone application (APP), which will be made available by the researchers, at the same time as the polysomnography exam.
Diagnostic Test: Polysomnography — All participants slept for one night in a sleep laboratory for PSG recording. The data will be confirmed by an otorhinolaryngology certified by the Brazilian Association of Sleep Disorders

SUMMARY:
Evaluate the correlation among the diagnostics of sleep bruxism and sleep quality obtained from the use of smartphone application (APP-Sleep Cycle®), PSG and questionnaires (Pittsburgh Sleep Quality Index-IQSP and Johansson).

DETAILED DESCRIPTION:
This study will evaluate the correlation between sleep bruxism and sleep quality diagnoses obtained using the application of the smartphone (APP-Sleep Cycle®), polysomnography and questionnaires (Pittsburgh Sleep Quality Index-IQSP and Johansson). Subjects (n = 40) between 19 and 60 years old will be submitted to polysomnography from January to December 2019. The questionnaires will be applied before the polysomnography, and the APP will be used together with the polysomnography. The data will be tabulated and a descriptive statistical analysis performed. Specific statistical tests will be determined after preliminary analysis of the data (α = 0.05).

ELIGIBILITY:
Inclusion Criteria:

* Adults (aged 20 to 60 years) and elderly (aged > 60 years) (WHO-World Health Organization, 2015) who will be undergone PSG at the Pelotas Sleep Institute (ISP);
* Adequate cognitive capacity to understand and answer the questionnaire.

Exclusion Criteria:

• Those which the participants were unable to answer the questionnaires and who presented a history of epilepsy that could interfere in the results of PSG.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All adults (aged 20 to 60 years) and elderly (aged > 60 years) who had undergone PSG at the Pelotas Sleep Institute (ISP), a private medical out patients clinic, from January to December 2019, will be invited to participate in the study.
  Eligibility criteria includ adequate cognitive capacity to understand and answer the questionnaire. Written consent will be given by all participants who agreed to participate in the study.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Data Collect on Sleep Quality with ISQP quastionario. | 4 months after study start
  Sleep quality data will be collected from the ISQP quastionario
Data Collect on Sleep Quality with the APP | 4 months after study start
  The sleep quality data will be collected in the APP along with the polysomnography exam, and the efficiency of the sleep is measured (god >80% or bad <80%).
Data Collect on Sleep Quality with polysomnography exam | 4 months after study start
  The sleep quality data will be collected in the polysomnography exam along with the APP, and the efficiency of the sleep is measured (god >80% or bad <80%).

CONTACTS AND LOCATIONS:
Overall Officials: Noéli Boscato, PhD, Principal Investigator — Federal University of Pelotas
Locations (1):
- Noéli Boscato, Pelotas, Rio Grande do Sul, Brazil